CLINICAL TRIAL: NCT01794923
Title: PLACEBO-CONTROLLED, DOUBLE-BLIND EVALUATION OF THE EFFICACY AND SAFETY OF IBUPROFEN 5% TOPICAL GEL FOR THE TREATMENT OF DELAYED-ONSET MUSCLE SORENESS OF THE ELBOW FLEXOR MUSCLES
Brief Title: Topical Ibuprofen for Delayed Onset Mulscle Soreness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3491010
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Pain
Keywords: Delayed onset muscle soreness; ibuprofen; topical
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ibuprofen 5% topical gel BID (Experimental): IBU BID (Treatment A)
  Interventions: Drug: IBU BID
- Placebo topical gel BID (Placebo Comparator): Placebo BID (Treatment B)
  Interventions: Drug: Placebo BID
- Ibuprofen 5% topical gel TID (Experimental): IBU TID (Treatment C)
  Interventions: Drug: IBU TID
- Placebo topical gel TID (Placebo Comparator): Placebo TID (Treatment D)
  Interventions: Drug: Placebo TID

INTERVENTIONS:
Drug: IBU BID — 10-cm strip of IBU 5% topical gel applied to the affected area BID (twice daily) x 3 days
  Arms: Ibuprofen 5% topical gel BID
Drug: Placebo BID — 10-cm strip of placebo topical gel applied to the affected area BID (twice daily) x 3 days
  Arms: Placebo topical gel BID
Drug: IBU TID — 10-cm strip of IBU 5% topical gel applied to the affected area TID (three times daily) x 3 days
  Arms: Ibuprofen 5% topical gel TID
Drug: Placebo TID — 10-cm strip of placebo topical gel applied to the affected area TID (three times daily) x 3 days
  Arms: Placebo topical gel TID

SUMMARY:
The objective of this study is to compare the efficacy and safety of Ibuprofen 5% Topical Gel versus placebo administered two or three times daily for the treatment of pain associated with delayed onset muscle soreness following intense eccentric exercise of the elbow flexor muscles.

ELIGIBILITY:
Inclusion Criteria:

Males or females, 18 to 65 years of age, who have not engaged in upper extremity fitness activities for a minimum of 3 months prior to entry in the study; subjects must be willing to refrain from use of pharmacologic or non pharmacologic treatments (ie, heat, ice, massage) and other forms of soreness relief during the study

Exclusion Criteria:

Use of corticosteroids or short- or long-acting non-steroidal anti-inflammatory drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2013-06-13 (Actual); Primary Completion 2014-03-29 (Actual); Study Completion 2014-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Institute for Applied Pharmaceutical Research, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3491010&StudyName=Topical%20Ibuprofen%20for%20Delayed%20Onset%20Mulscle%20Soreness

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Combined: Placebo matched to Ibuprofen topical gel applied topically as a 4 inch strip twice daily (to match Ibuprofen twice daily regimen) or three times daily (to match Ibuprofen thrice daily regimen) on Days 1, 2 and 3.
- Ibuprofen Twice Daily: Ibuprofen 5 percent (%) topical gel applied topically as a 4-inch strip twice daily on Day 1, 2 and 3.
- Ibuprofen Three Times Daily: Ibuprofen 5% topical gel applied topically as a 4 inch strip three times daily on Day 1, 2 and 3.
Period: Overall Study
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Started | 83 | 60 | 62
Completed | 83 | 60 | 61
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily | Total
Number analyzed (Participants) | 83 | 60 | 62 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (14.79) | 44.4 (13.19) | 45.5 (13.08) | 43.4 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 41 | 41 | 137
  Male | 28 | 19 | 21 | 68
Muscle Soreness with Movement (MSM) [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to complete one preacher curl, using the arm that was exercised earlier to stimulate muscle soreness on movement. Upon completion of preacher curl, participants were asked to rate their degree of muscle soreness with movement, using an 11-point scale ranging from 0 to 10, where 0 signifies 'not sore' and 10 signifies 'extremely sore', higher score= more severity.
  units on a scale | 7.7 (1.21) | 7.6 (1.09) | 7.4 (1.11) | 7.6 (1.15)
Stiffness during Muscle Soreness with Movement (SMSM) [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to rate their stiffness during muscle soreness with movement, using an 11-point scale, with 0 = 'not stiff' and 10 = 'extremely stiff', higher score= more severity.
  units on a scale | 7.5 (1.32) | 7.6 (1.18) | 7.4 (1.28) | 7.5 (1.26)
Spontaneous Muscle Soreness (SMS) [Mean (Standard Deviation); unit: units on a scale] — Participants after sitting quietly for 3 minutes, were asked to extend the arm which was exercised earlier to stimulate muscle soreness on movement. Participants were asked to rate their degree of spontaneous muscle soreness, using an 11-point scale ranging from 0 to 10, where 0 signifies 'not sore' and 10 signifies 'extremely sore', higher score=more severity.
  units on a scale | 7.1 (1.16) | 7.1 (1.13) | 7.3 (1.16) | 7.2 (1.15)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Time-Weighted Sum of Muscle Soreness With Movement Over 0-24 Hours Post-Dose 1 (MSM 0-24 )
Description: Participants were asked to complete one preacher curl, using the arm that was exercised earlier to stimulate muscle soreness on movement (MSM). Upon completion of preacher curl, participants were asked to rate their degree of MSM, using an 11 point scale ranging from 0 to 10, where 0=not sore and 10=extremely sore, higher score=more severity. Change from baseline in the time-weighted sum of MSM over 0-24 hours was derived as the MSM change from baseline multiplied by time elapsed since the previous assessment and summed over all assessments from Hour 0 to Hour 24 (range: -96 to 240, higher score indicates better response).
Time Frame: Baseline, 0 to 24 hours post-Dose 1 on Day 1
Population: Full analysis set population included all randomized participants who were dosed with the study medication and provided a baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 83 | 60 | 62
units on a scale | 22.2 (4.46) | 17.8 (5.12) | 29.7 (5.00)
Statistical Analysis 1: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; Analysis was performed using an analysis of variance (ANOVA) model with treatment, baseline categorical pain severity rating (PSR), sex, and baseline muscle soreness with movement (MSM) terms; Test type: Superiority or Other; p = 0.200, ANOVA
Statistical Analysis 2: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; Analysis was performed using an ANOVA model with treatment, baseline categorical pain severity rating (PSR), sex, and baseline muscle soreness with movement (MSM) terms; Test type: Superiority or Other; p = 0.230, ANOVA; Least Squares (LS) Mean Difference = 7.6, 95% CI 2-sided [-4.81 to 19.92]
Statistical Analysis 3: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.484, ANOVA; LS Mean Difference = -4.4, 95% CI 2-sided [-16.81 to 7.99]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.077, ANOVA; LS Mean Difference = 12.0, 95% CI 2-sided [-1.32 to 25.25]

2. Secondary Outcome: Change From Baseline in the Time-Weighted Sum of Muscle Soreness With Movement Over 24-48 Hours, 48-72 Hours, 0-72 Hours Post-Dose 1
Description: Participants were asked to complete one preacher curl, using the arm that was exercised earlier to stimulate MSM. Upon completion of preacher curl, participants were asked to rate their degree of MSM, using an 11-point scale ranging from 0 to 10, where 0=not sore and 10=extremely sore, higher scores=more severity. Change from baseline in the time-weighted sum of MSM over 24-48 hours, 48-72 hours and 0-72 hours were derived as the MSM change from baseline multiplied by time elapsed since the previous assessment and summed over all assessments from Hour 24 to Hour 48 (range: -96 to 240, higher score indicates better response); Hour 48 to Hour 72 (range: -96 to 240, higher score indicates better outcome); and Hour 0 to Hour 72 (range: -288 to 720, higher score indicates better response).
Time Frame: Baseline, 24 to 48, 48 to 72, 0 to 72 hours post-Dose 1 on Day 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 83 | 60 | 62
units on a scale
  28-48 hours | 78.3 (9.14) | 81.0 (10.49) | 85.4 (10.25)
  48-72 hours | 149.6 (10.06) | 150.5 (11.54) | 135.6 (11.27)
  0-72 hours | 194.6 (16.26) | 191.9 (18.66) | 191.4 (18.22)
Statistical Analysis 1: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 24-48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.860, ANOVA
Statistical Analysis 2: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.584, ANOVA; LS Mean Difference = 7.0, 95% CI 2-sided [-18.30 to 32.38]
Statistical Analysis 3: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.838, ANOVA; LS Mean Difference = 2.6, 95% CI 2-sided [-22.77 to 28.06]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.750, ANOVA; LS Mean Difference = 4.4, 95% CI 2-sided [-22.81 to 31.61]
Statistical Analysis 5: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 48-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.533, ANOVA
Statistical Analysis 6: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.326, ANOVA; LS Mean Difference = -13.9, 95% CI 2-sided [-41.81 to 13.95]
Statistical Analysis 7: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.945, ANOVA; LS Mean Difference = 1.0, 95% CI 2-sided [-26.98 to 28.94]
Statistical Analysis 8: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.327, ANOVA; LS Mean Difference = -14.9, 95% CI 2-sided [-44.85 to 15.03]
Statistical Analysis 9: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 0-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.988, ANOVA
Statistical Analysis 10: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.887, ANOVA; LS Mean Difference = -3.2, 95% CI 2-sided [-48.31 to 41.81]
Statistical Analysis 11: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.907, ANOVA; LS Mean Difference = -2.7, 95% CI 2-sided [-47.88 to 42.50]
Statistical Analysis 12: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 2, analysis 9]; Test type: Superiority or Other; p = 0.982, ANOVA; LS Mean Difference = -0.6, 95% CI 2-sided [-48.95 to 47.83]

3. Secondary Outcome: Change From Baseline in Muscle Soreness With Movement at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 24, 30, 36, 48, 54, 60 and 72 Hours Post-Dose 1
Description: Participants were asked to complete one preacher curl, using the arm that was exercised earlier to stimulate MSM. Upon completion of preacher curl, participants were asked to rate their degree of MSM, using an 11-point scale ranging from 0 to 10, where 0=not sore' and 10=extremely sore, higher score=more severity.
Time Frame: Baseline,1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 24, 30, 36, 48, 54, 60 and 72 hours post-Dose 1 on Day 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 83 | 60 | 62
units on a scale
  1 hour | -0.0 (0.10) | -0.1 (0.11) | -0.2 (0.11)
  2 hours | 0.1 (0.11) | -0.2 (0.12) | -0.0 (0.12)
  3 hours | 0.2 (0.13) | -0.1 (0.15) | 0.1 (0.15)
  4 hours | 0.4 (0.16) | 0.0 (0.18) | 0.2 (0.18)
  5 hours | 0.5 (0.16) | 0.1 (0.19) | 0.3 (0.18)
  6 hours | 0.5 (0.18) | 0.2 (0.21) | 0.5 (0.21)
  7 hours | 0.7 (0.19) | 0.3 (0.22) | 0.7 (0.22)
  8 hours | 0.7 (0.20) | 0.4 (0.23) | 0.7 (0.22)
  9 hours | 0.7 (0.21) | 0.3 (0.24) | 0.1 (0.23)
  10 hours | 0.9 (0.21) | 0.5 (0.25) | 1.1 (0.24)
  11 hours | 0.8 (0.21) | 0.5 (0.24) | 1.1 (0.23)
  12 hours | 0.9 (0.22) | 0.6 (0.25) | 1.2 (0.25)
  24 hours | 1.3 (0.26) | 1.3 (0.29) | 1.9 (0.29)
  30 hours | 1.7 (0.26) | 1.7 (0.30) | 2.0 (0.29)
  36 hours | 2.1 (0.28) | 2.2 (0.33) | 2.3 (0.32)
  48 hours | 3.3 (0.29) | 3.5 (0.33) | 3.0 (0.33)
  54 hours | 3.7 (0.30) | 3.6 (0.34) | 3.5 (0.33)
  60 hours | 4.2 (0.30) | 4.2 (0.34) | 3.9 (0.33)
  72 hours | 5.2 (0.29) | 5.1 (0.33) | 4.6 (0.32)
Statistical Analysis 1: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 1 Hour: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.630, ANOVA
Statistical Analysis 2: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.342, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.39 to 0.14]
Statistical Analysis 3: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.600, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.34 to 0.19]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.691, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.34 to 0.23]
Statistical Analysis 5: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 2 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.091, ANOVA
Statistical Analysis 6: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.351, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.44 to 0.16]
Statistical Analysis 7: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.029, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.64 to -0.04]
Statistical Analysis 8: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.238, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.13 to 0.52]
Statistical Analysis 9: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 3 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.305, ANOVA
Statistical Analysis 10: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; p = 0.370, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.54 to 0.20]
Statistical Analysis 11: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; p = 0.130, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.66 to 0.09]
Statistical Analysis 12: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; p = 0.561, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.28 to 0.51]
Statistical Analysis 13: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 4 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.209, ANOVA
Statistical Analysis 14: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; p = 0.277, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.68 to 0.19]
Statistical Analysis 15: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; p = 0.085, ANOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-0.82 to 0.05]
Statistical Analysis 16: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 13]; Test type: Superiority or Other; p = 0.546, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.32 to 0.61]
Statistical Analysis 17: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 5 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.185, ANOVA
Statistical Analysis 18: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; p = 0.400, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.64 to 0.26]
Statistical Analysis 19: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; p = 0.067, ANOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-0.88 to 0.03]
Statistical Analysis 20: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 17]; Test type: Superiority or Other; p = 0.350, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.25 to 0.71]
Statistical Analysis 21: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 6 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.493, ANOVA
Statistical Analysis 22: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.922, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.53 to 0.48]
Statistical Analysis 23: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.265, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.80 to 0.22]
Statistical Analysis 24: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.342, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.28 to 0.81]
Statistical Analysis 25: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 7 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.311, ANOVA
Statistical Analysis 26: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; p = 0.865, ANOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.49 to 0.58]
Statistical Analysis 27: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; p = 0.193, ANOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-0.89 to 0.18]
Statistical Analysis 28: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; p = 0.170, ANOVA; LS Mean Difference = 0.4, 95% CI 2-sided [-0.17 to 0.97]
Statistical Analysis 29: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 8 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.383, ANOVA
Statistical Analysis 30: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; p = 0.802, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.48 to 0.62]
Statistical Analysis 31: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; p = 0.260, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.87 to 0.24]
Statistical Analysis 32: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; p = 0.199, ANOVA; LS Mean Difference = 0.4, 95% CI 2-sided [-0.21 to 0.98]
Statistical Analysis 33: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 9 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.139, ANOVA
Statistical Analysis 34: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; p = 0.441, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.35 to 0.80]
Statistical Analysis 35: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; p = 0.183, ANOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-0.96 to 0.18]
Statistical Analysis 36: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; p = 0.050, ANOVA; LS Mean Difference = 0.6, 95% CI 2-sided [-0.00 to 1.23]
Statistical Analysis 37: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 10 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.221, ANOVA
Statistical Analysis 38: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 37]; Test type: Superiority or Other; p = 0.526, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.40 to 0.79]
Statistical Analysis 39: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 37]; Test type: Superiority or Other; p = 0.232, ANOVA; LS mean Difference = -0.4, 95% CI 2-sided [-0.96 to 0.23]
Statistical Analysis 40: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 37]; Test type: Superiority or Other; p = 0.089, ANOVA; LS Mean Difference = 0.6, 95% CI 2-sided [-0.08 to 1.19]
Statistical Analysis 41: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 11 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.190, ANOVA
Statistical Analysis 42: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; p = 0.365, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.31 to 0.85]
Statistical Analysis 43: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; p = 0.295, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.89 to 0.27]
Statistical Analysis 44: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; p = 0.069, ANOVA; LS Mean Difference = 0.6, 95% CI 2-sided [-0.05 to 1.20]
Statistical Analysis 45: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 12 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.197, ANOVA
Statistical Analysis 46: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 45]; Test type: Superiority or Other; p = 0.309, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.29 to 0.92]
Statistical Analysis 47: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 45]; Test type: Superiority or Other; p = 0.359, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.89 to 0.33]
Statistical Analysis 48: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 45]; Test type: Superiority or Other; p = 0.072, ANOVA; LS Mean Difference = 0.6, 95% CI 2-sided [-0.05 to 1.25]
Statistical Analysis 49: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.151, ANOVA
Statistical Analysis 50: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 49]; Test type: Superiority or Other; p = 0.090, ANOVA; LS Mean Difference = 0.6, 95% CI 2-sided [-0.10 to 1.32]
Statistical Analysis 51: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 49]; Test type: Superiority or Other; p = 0.889, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.76 to 0.66]
Statistical Analysis 52: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 49]; Test type: Superiority or Other; p = 0.088, ANOVA; LS Mean Difference = 0.7, 95% CI 2-sided [-0.10 to 1.42]
Statistical Analysis 53: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 30 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.673, ANOVA
Statistical Analysis 54: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 53]; Test type: Superiority or Other; p = 0.393, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.41 to 1.04]
Statistical Analysis 55: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 53]; Test type: Superiority or Other; p = 0.887, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.67 to 0.78]
Statistical Analysis 56: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 53]; Test type: Superiority or Other; p = 0.507, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.51 to 1.04]
Statistical Analysis 57: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 36 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.873, ANOVA
Statistical Analysis 58: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 57]; Test type: Superiority or Other; p = 0.605, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.58 to 1.00]
Statistical Analysis 59: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 26 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.860, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.72 to 0.86]
Statistical Analysis 60: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 57]; Test type: Superiority or Other; p = 0.751, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.71 to 0.98]
Statistical Analysis 61: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.528, ANOVA
Statistical Analysis 62: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 61]; Test type: Superiority or Other; p = 0.486, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-1.09 to 0.52]
Statistical Analysis 63: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 61]; Test type: Superiority or Other; p = 0.610, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.60 to 1.02]
Statistical Analysis 64: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 61]; Test type: Superiority or Other; p = 0.261, ANOVA; LS Mean Difference = -0.5, 95% CI 2-sided [-1.36 to 0.37]
Statistical Analysis 65: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 54 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.943, ANOVA
Statistical Analysis 66: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 65]; Test type: Superiority or Other; p = 0.733, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.96 to 0.68]
Statistical Analysis 67: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 65]; Test type: Superiority or Other; p = 0.902, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.87 to 0.77]
Statistical Analysis 68: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 65]; Test type: Superiority or Other; p = 0.840, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.97 to 0.79]
Statistical Analysis 69: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 60 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.758, ANOVA
Statistical Analysis 70: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 69]; Test type: Superiority or Other; p = 0.493, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-1.12 to 0.54]
Statistical Analysis 71: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 69]; Test type: Superiority or Other; p = 0.974, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.84 to 0.82]
Statistical Analysis 72: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 69]; Test type: Superiority or Other; p = 0.543, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-1.16 to 0.61]
Statistical Analysis 73: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.238, ANOVA
Statistical Analysis 74: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 73]; Test type: Superiority or Other; p = 0.106, ANOVA; LS Mean Difference = -0.7, 95% CI 2-sided [-1.46 to 0.14]
Statistical Analysis 75: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 3, analysis 73]; Test type: Superiority or Other; p = 0.817, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.90 to 0.71]
Statistical Analysis 76: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 3, analysis 73]; Test type: Superiority or Other; p = 0.197, ANOVA; LS Mean Difference = -0.6, 95% CI 2-sided [-1.43 to 0.30]

4. Secondary Outcome: Change From Baseline in the Time-weighted Sum of Spontaneous Muscle Soreness Over 0-24 Hours, 24-48 Hours, 48-72 Hours, and 0-72 Hours Post-Dose 1
Description: Participants after sitting quietly for 3 minutes, were asked to extend the arm that was exercised earlier to stimulate MSM. Participants were asked to rate their degree of SMS, using an 11-point scale ranging from 0 to 10, where 0=not sore and 10=extremely sore, higher score=more severity. Change from baseline in time-weighted sum of SMS over 0-24 hours (hr.), 24-48 hr., 48-72 hr. and 0-72 hr. were derived as the SMS change from baseline multiplied by time elapsed since the previous assessment and summed overall assessment from Hour 0 to Hour 24 (range: -240 to 240, higher score indicates better response), Hour 24 to Hour 48 (range: -240 to 240, higher score indicates better response); Hour 48 to Hour 72 (range: -240 to 240, higher score indicates better response); and Hour 0 to Hour 72 (range: -720 to 720, higher score indicates better response).
Time Frame: Baseline, 24 to 48, 48 to 72, 0 to 72 hours post-Dose 1 on Day 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 83 | 60 | 62
units on a scale
  0-24 hours | 21.8 (4.50) | 18.7 (5.23) | 24.6 (5.37)
  24-48 hours | 77.3 (8.95) | 78.0 (10.41) | 73.1 (10.69)
  48-72 hours | 143.9 (9.64) | 146.0 (11.20) | 124.9 (11.50)
  0-72 hours | 188.7 (15.83) | 187.7 (18.40) | 170.8 (18.89)
Statistical Analysis 1: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 0-24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline spontaneous muscle soreness (SMS) terms; Test type: Superiority or Other; p = 0.702, ANOVA
Statistical Analysis 2: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.664, ANOVA; LS Mean Difference = 2.8, 95% CI 2-sided [-9.91 to 15.53]
Statistical Analysis 3: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.637, ANOVA; LS Mean Difference = -3.0, 95% CI 2-sided [-15.77 to 9.68]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 0-24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline MSM terms; Test type: Superiority or Other; p = 0.401, ANOVA; LS Mean Difference = 5.9, 95% CI 2-sided [-7.85 to 19.57]
Statistical Analysis 5: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 24-48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline spontaneous muscle soreness (SMS) terms; Test type: Superiority or Other; p = 0.926, ANOVA
Statistical Analysis 6: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.743, ANOVA; LS Mean Difference = -4.2, 95% CI 2-sided [-29.51 to 21.10]
Statistical Analysis 7: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.952, ANOVA; LS Mean Difference = 0.8, 95% CI 2-sided [-24.55 to 26.08]
Statistical Analysis 8: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.719, ANOVA; LS Mean Difference = -5.0, 95% CI 2-sided [-32.25 to 22.30]
Statistical Analysis 9: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 48-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline spontaneous muscle soreness (SMS) terms; Test type: Superiority or Other; p = 0.284, ANOVA
Statistical Analysis 10: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.171, ANOVA; LS Mean Difference = -19.0, 95% CI 2-sided [-46.21 to 8.28]
Statistical Analysis 11: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.875, ANOVA; LS Mean Difference = 2.2, 95% CI 2-sided [-25.08 to 29.42]
Statistical Analysis 12: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.157, ANOVA; LS Mean Difference = -21.1, 95% CI 2-sided [-50.50 to 8.23]
Statistical Analysis 13: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 0-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline spontaneous muscle soreness (SMS) terms; Test type: Superiority or Other; p = 0.699, ANOVA
Statistical Analysis 14: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.433, ANOVA; LS Mean Difference = -17.8, 95% CI 2-sided [-62.58 to 26.90]
Statistical Analysis 15: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.966, ANOVA; LS Mean Difference = -1.0, 95% CI 2-sided [-45.73 to 43.78]
Statistical Analysis 16: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 4, analysis 13]; Test type: Superiority or Other; p = 0.491, ANOVA; LS Mean Difference = -16.9, 95% CI 2-sided [-65.08 to 31.36]

5. Secondary Outcome: Change From Baseline in Spontaneous Muscle Soreness at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 24, 30, 36, 48, 54, 60 and 72 Hours Post-Dose 1
Description: Participants after sitting quietly for 3 minutes, were asked to extend the arm that was exercised earlier to stimulate SMS. Participants were asked to rate their degree of SMS, using an 11-point scale ranging from 0 to 10, where 0=not sore and 10=extremely sore, higher score=more severity.
Time Frame: Baseline,1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 24, 30, 36, 48, 54, 60 and 72 hours post-Dose 1 on Day 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 83 | 60 | 62
units on a scale
  1 hour | 0.0 (0.08) | 0.1 (0.09) | -0.1 (0.10)
  2 hours | 0.1 (0.10) | -0.0 (0.11) | -0.2 (0.12)
  3 hours | 0.2 (0.13) | 0.1 (0.15) | -0.1 (0.16)
  4 hours | 0.4 (0.15) | 0.2 (0.17) | 0.1 (0.18)
  5 hours | 0.4 (0.17) | 0.2 (0.19) | 0.3 (0.20)
  6 hours | 0.5 (0.18) | 0.3 (0.21) | 0.4 (0.22)
  7 hours | 0.7 (0.19) | 0.4 (0.22) | 0.7 (0.23)
  8 hours | 0.8 (0.20) | 0.5 (0.23) | 0.8 (0.24)
  9 hours | 0.8 (0.21) | 0.6 (0.24) | 1.0 (0.25)
  10 hours | 0.9 (0.21) | 0.6 (0.24) | 1.0 (0.25)
  11 hours | 0.9 (0.22) | 0.6 (0.25) | 1.1 (0.26)
  12 hours | 0.9 (0.22) | 0.7 (0.25) | 1.2 (0.26)
  24 hours | 1.3 (0.26) | 1.2 (0.30) | 1.5 (031)
  30 hours | 1.7 (0.26) | 1.7 (0.30) | 1.6 (0.31)
  36 hours | 2.2 (0.28) | 2.1 (0.32) | 1.9 (0.33)
  48 hours | 3.2 (0.28) | 3.4 (0.32) | 2.8 (0.33)
  54 hours | 3.7 (0.29) | 3.6 (0.33) | 3.2 (0.34)
  60 hours | 4.0 (0.29) | 4.1 (0.33) | 3.5 (0.34)
  72 hours | 4.9 (0.28) | 4.9 (0.32) | 4.3 (0.33)
Statistical Analysis 1: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 1 Hour: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.219, ANOVA
Statistical Analysis 2: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.214, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.37 to 0.08]
Statistical Analysis 3: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.555, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.16 to 0.29]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.090, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.45 to 0.03]
Statistical Analysis 5: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 2 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.161, ANOVA
Statistical Analysis 6: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.056, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.55 to 0.01]
Statistical Analysis 7: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.395, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.40 to 0.16]
Statistical Analysis 8: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.324, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.45 to 0.15]
Statistical Analysis 9: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 3 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.246, ANOVA
Statistical Analysis 10: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 9]; Test type: Superiority or Other; p = 0.094, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.68 to 0.05]
Statistical Analysis 11: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 9]; Test type: Superiority or Other; p = 0.491, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.50 to 0.24]
Statistical Analysis 12: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 9]; Test type: Superiority or Other; p = 0.359, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.58 to 0.21]
Statistical Analysis 13: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 4 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.294, ANOVA
Statistical Analysis 14: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.136, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.74 to 0.10]
Statistical Analysis 15: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.293, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.65 to 0.20]
Statistical Analysis 16: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.682, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.55 to 0.36]
Statistical Analysis 17: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 5 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.747, ANOVA
Statistical Analysis 18: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 17]; Test type: Superiority or Other; p = 0.592, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.60 to 0.34]
Statistical Analysis 19: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 17]; Test type: Superiority or Other; p = 0.473, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.64 to 0.30]
Statistical Analysis 20: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 17]; Test type: Superiority or Other; p = 0.866, ANOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.46 to 0.55]
Statistical Analysis 21: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 6 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.776, ANOVA
Statistical Analysis 22: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.761, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.59 to 0.43]
Statistical Analysis 23: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.477, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.69 to 0.33]
Statistical Analysis 24: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 21]; Test type: Superiority or Other; p = 0.705, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.44 to 0.65]
Statistical Analysis 25: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 7 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.600, ANOVA
Statistical Analysis 26: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 25]; Test type: Superiority or Other; p = 0.931, ANOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.52 to 0.56]
Statistical Analysis 27: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 25]; Test type: Superiority or Other; p = 0.381, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.78 to 0.30]
Statistical Analysis 28: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 25]; Test type: Superiority or Other; p = 0.371, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.32 to 0.85]
Statistical Analysis 29: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 8 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.670, ANOVA
Statistical Analysis 30: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 29]; Test type: Superiority or Other; p = 0.941, ANOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.54 to 0.58]
Statistical Analysis 31: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 29]; Test type: Superiority or Other; p = 0.437, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.78 to 0.34]
Statistical Analysis 32: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 29]; Test type: Superiority or Other; p = 0.429, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.36 to 0.84]
Statistical Analysis 33: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 9 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.484, ANOVA
Statistical Analysis 34: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 33]; Test type: Superiority or Other; p = 0.504, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.38 to 0.78]
Statistical Analysis 35: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 33]; Test type: Superiority or Other; p = 0.528, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.77 to 0.40]
Statistical Analysis 36: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 33]; Test type: Superiority or Other; p = 0.229, ANOVA; LS Mean Difference = 0.4, 95% CI 2-sided [-0.24 to 1.01]
Statistical Analysis 37: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 10 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.536, ANOVA
Statistical Analysis 38: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 37]; Test type: Superiority or Other; p = 0.728, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.49 to 0.70]
Statistical Analysis 39: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 37]; Test type: Superiority or Other; p = 0.414, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.84 to 0.35]
Statistical Analysis 40: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 37]; Test type: Superiority or Other; p = 0.280, ANOVA; LS Mean Difference = 0.4, 95% CI 2-sided [-0.29 to 0.99]
Statistical Analysis 41: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 11 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.402, ANOVA
Statistical Analysis 42: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 41]; Test type: Superiority or Other; p = 0.513, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.41 to 0.81]
Statistical Analysis 43: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 41]; Test type: Superiority or Other; p = 0.424, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.86 to 0.36]
Statistical Analysis 44: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 41]; Test type: Superiority or Other; p = 0.178, ANOVA; LS Mean Difference = 0.4, 95% CI 2-sided [-0.21 to 1.10]
Statistical Analysis 45: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 12 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.442, ANOVA
Statistical Analysis 46: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 45]; Test type: Superiority or Other; p = 0.357, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.33 to 0.91]
Statistical Analysis 47: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 45]; Test type: Superiority or Other; p = 0.675, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.75 to 0.49]
Statistical Analysis 48: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 45]; Test type: Superiority or Other; p = 0.215, ANOVA; LS Mean Difference = 0.4, 95% CI 2-sided [-0.25 to 1.09]
Statistical Analysis 49: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.643, ANOVA
Statistical Analysis 50: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 49]; Test type: Superiority or Other; p = 0.466, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.46 to 0.99]
Statistical Analysis 51: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 49]; Test type: Superiority or Other; p = 0.818, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.81 to 0.64]
Statistical Analysis 52: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 49]; Test type: Superiority or Other; p = 0.373, ANOVA; LS Mean Difference = 0.4, 95% CI 2-sided [-0.43 to 1.13]
Statistical Analysis 53: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 30 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.984, ANOVA
Statistical Analysis 54: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 53]; Test type: Superiority or Other; p = 0.874, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.79 to 0.68]
Statistical Analysis 55: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 53]; Test type: Superiority or Other; p = 0.990, ANOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.73 to 0.74]
Statistical Analysis 56: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 53]; Test type: Superiority or Other; p = 0.875, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.85 to 0.73]
Statistical Analysis 57: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 36 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.841, ANOVA
Statistical Analysis 58: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 57]; Test type: Superiority or Other; p = 0.580, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-1.01 to 0.57]
Statistical Analysis 59: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 57]; Test type: Superiority or Other; p = 0.958, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.81 to 0.77]
Statistical Analysis 60: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 57]; Test type: Superiority or Other; p = 0.643, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-1.05 to 0.65]
Statistical Analysis 61: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.299, ANOVA
Statistical Analysis 62: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 61]; Test type: Superiority or Other; p = 0.230, ANOVA; LS mean Difference = -0.5, 95% CI 2-sided [-1.26 to 0.31]
Statistical Analysis 63: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 61]; Test type: Superiority or Other; p = 0.694, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.63 to 0.94]
Statistical Analysis 64: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 61]; Test type: Superiority or Other; p = 0.140, ANOVA; LS Mean Difference = -0.6, 95% CI 2-sided [-1.48 to 0.21]
Statistical Analysis 65: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 54 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.503, ANOVA
Statistical Analysis 66: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.262, ANOVA; LS Mean Difference = -0.5, 95% CI 2-sided [-1.28 to 0.35]
Statistical Analysis 67: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.871, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.88 to 0.75]
Statistical Analysis 68: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 65]; Test type: Superiority or Other; p = 0.373, ANOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-1.27 to 0.48]
Statistical Analysis 69: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 60 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.413, ANOVA
Statistical Analysis 70: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 69]; Test type: Superiority or Other; p = 0.317, ANOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-1.22 to 0.40]
Statistical Analysis 71: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 69]; Test type: Superiority or Other; p = 0.708, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.66 to 0.97]
Statistical Analysis 72: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 69]; Test type: Superiority or Other; p = 0.202, ANOVA; LS Mean Difference = -0.6, 95% CI 2-sided [-1.44 to 0.31]
Statistical Analysis 73: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMS terms; Test type: Superiority or Other; p = 0.190, ANOVA
Statistical Analysis 74: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 73]; Test type: Superiority or Other; p = 0.094, ANOVA; LS Mean Difference = -0.7, 95% CI 2-sided [-1.44 to 0.11]
Statistical Analysis 75: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 5, analysis 73]; Test type: Superiority or Other; p = 0.960, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.80 to 0.76]
Statistical Analysis 76: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 5, analysis 73]; Test type: Superiority or Other; p = 0.132, ANOVA; LS Mean Difference = -0.6, 95% CI 2-sided [-1.48 to 0.20]

6. Secondary Outcome: Time-weighted Sum of Muscle Soreness Relief Over 0-24 Hours, 24-48 Hours, 48-72 Hours, and 0-72 Hours
Description: Participants were asked: "Which phrase best describes the relief of muscle soreness which you are experiencing?" Participant's response were recorded using a five-point scale: 0=None, 1=A little, 2=Some, 3=A lot and 4=Complete relief. Time-weighted sum of muscle soreness relief over 0-24 hours, 24-48 hours, 48-72 hours, and 0-72 hours were derived as the muscle soreness relief score multiplied by time elapsed since the previous assessment and summed over all assessments from Hour 0 to Hour 24 (total score range: 0 [none] to 96 [complete relief], higher score indicates better response), Hour 24 to Hour 48 (range: 0 to 96, higher score indicates better response); Hour 48 to Hour 72 (range: 0 to 96, higher score indicates better response); and Hour 0 to Hour 72 (range: 0 to 288, higher score indicates better response).
Time Frame: 0 to 24, 24 to 48, 48 to 72 and 0 to 72 hours on Day 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 83 | 60 | 62
units on a scale
  0-24 hours | 18.8 (2.26) | 16.8 (2.64) | 23.4 (2.61)
  24-48 hours | 57.3 (4.31) | 56.4 (5.04) | 58.4 (4.98)
  48-72 hours | 90.5 (4.19) | 92.5 (4.89) | 82.3 (4.83)
  0-72 hours | 128.6 (7.18) | 127.2 (8.39) | 124.4 (8.29)
Statistical Analysis 1: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 0-24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.163, ANOVA
Statistical Analysis 2: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 0-24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.162, ANOVA; LS Mean Difference = 4.6, 95% CI 2-sided [-1.86 to 11.02]
Statistical Analysis 3: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 0-24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.559, ANOVA; LS Mean Difference = -1.9, 95% CI 2-sided [-8.42 to 4.57]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 0-24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.066, ANOVA; LS Mean Difference = 6.5, 95% CI 2-sided [-0.44 to 13.45]
Statistical Analysis 5: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 24-48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.957, ANOVA
Statistical Analysis 6: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 24-48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.864, ANOVA; LS Mean Difference = 1.1, 95% CI 2-sided [-11.20 to 13.33]
Statistical Analysis 7: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 24-48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.883, ANOVA; LS Mean Difference = -0.9, 95% CI 2-sided [-13.30 to 11.45]
Statistical Analysis 8: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 24-48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.767, ANOVA; LS Mean Difference = 2.0, 95% CI 2-sided [-11.24 to 15.22]
Statistical Analysis 9: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 48-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.243, ANOVA
Statistical Analysis 10: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 48-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.176, ANOVA; LS Mean Difference = -8.2, 95% CI 2-sided [-20.12 to 3.70]
Statistical Analysis 11: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 48-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.741, ANOVA; LS Mean Difference = 2.0, 95% CI 2-sided [-10.00 to 14.03]
Statistical Analysis 12: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 48-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.118, ANOVA; LS Mean Difference = -10.2, 95% CI 2-sided [-23.07 to 2.62]
Statistical Analysis 13: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 0-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.920, ANOVA
Statistical Analysis 14: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 0-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.685, ANOVA; LS Mean Difference = -4.2, 95% CI 2-sided [-24.64 to 16.23]
Statistical Analysis 15: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 0-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.892, ANOVA; LS Mean Difference = -1.4, 95% CI 2-sided [-22.04 to 19.19]
Statistical Analysis 16: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 0-72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.804, ANOVA; LS Mean Difference = -2.8, 95% CI 2-sided [-24.82 to 19.25]

7. Secondary Outcome: Change From Baseline in Stiffness During Muscle Soreness With Movement (SMSM) Assessment at 24 Hours Post-Dose 1
Description: Participants were asked to rate their SMSM, using an 11-point scale, with 0=not stiff and 10=extremely stiff, higher score indicated more severity.
Time Frame: Baseline, 24 hours post-Dose 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 83 | 60 | 62
units on a scale | 1.6 (0.31) | 1.7 (0.37) | 2.1 (0.36)
Statistical Analysis 1: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMSM terms; Test type: Superiority or Other; p = 0.533, ANOVA
Statistical Analysis 2: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMSM terms; Test type: Superiority or Other; p = 0.266, ANOVA; LS Mean Difference = 0.5, 95% CI 2-sided [-0.38 to 1.38]
Statistical Analysis 3: Comparison: Placebo Combined vs Ibuprofen Twice Daily; Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMSM terms; Test type: Superiority or Other; p = 0.730, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.74 to 1.05]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; Analysis was performed using an ANOVA model with treatment, baseline categorical PSR, sex, and baseline SMSM terms; Test type: Superiority or Other; p = 0.479, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.61 to 1.30]

8. Secondary Outcome: Muscle Soreness Relief at Each Time Point
Description: Participants were asked: "Which phrase best describes the relief of muscle soreness which you are experiencing?" Participant's response was recorded using a five-point scale: 0 = None, 1 = A little, 2 = Some, 3 = A lot and 4 = Complete, higher scores indicated better response/more relief.
Time Frame: 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 24, 30, 36, 48, 54, 60 and 72 hours post-Dose 1 on Day 1
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 83 | 60 | 62
units on a scale
  1 hour | 0.1 (0.04) | 0.1 (0.05) | 0.0 (0.05)
  2 hours | 0.2 (0.05) | 0.2 (0.05) | 0.2 (0.05)
  3 hours | 0.3 (0.07) | 0.2 (0.08) | 0.3 (0.08)
  4 hours | 0.5 (0.08) | 0.4 (0.10) | 0.4 (0.10)
  5 hours | 0.5 (0.08) | 0.3 (0.10) | 0.5 (0.10)
  6 hours | 0.5 (0.10) | 0.5 (0.11) | 0.7 (0.11)
  7 hours | 0.6 (0.10) | 0.5 (0.11) | 0.7 (0.11)
  8 hours | 0.6 (0.10) | 0.6 (0.12) | 0.7 (0.12)
  9 hours | 0.7 (0.10) | 0.6 (0.12) | 0.9 (0.12)
  10 hours | 0.7 (0.11) | 0.7 (0.13) | 1.0 (0.13)
  11 hours | 0.7 (0.11) | 0.7 (0.13) | 1.0 (0.13)
  12 hours | 0.7 (0.11) | 0.7 (0.13) | 1.0 (0.13)
  24 hours | 1.0 (0.14) | 0.9 (0.16) | 1.3 (0.16)
  30 hours | 1.4 (0.14) | 1.3 (0.16) | 1.4 (0.16)
  36 hours | 1.8 (0.14) | 1.6 (0.16) | 1.7 (0.16)
  48 hours | 2.1 (0.13) | 2.3 (0.15) | 2.0 (0.15)
  54 hours | 2.4 (0.13) | 2.3 (0.15) | 2.2 (0.15)
  60 hours | 2.6 (0.13) | 2.5 (0.15) | 2.4 (0.15)
  72 hours | 2.9 (0.13) | 3.0 (0.15) | 2.6 (0.15)
Statistical Analysis 1: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 1 Hour: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.189, ANOVA
Statistical Analysis 2: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 1 Hour: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.389, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.17 to 0.07]
Statistical Analysis 3: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 1 Hour: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.273, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.05 to 0.19]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 1 Hour: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.069, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.25 to 0.01]
Statistical Analysis 5: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 2 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.716, ANOVA
Statistical Analysis 6: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 2 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.735, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.15 to 0.11]
Statistical Analysis 7: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 2 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.414, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.19 to 0.08]
Statistical Analysis 8: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 2 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.652, ANOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.11 to 0.17]
Statistical Analysis 9: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 3 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.622, ANOVA
Statistical Analysis 10: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 3 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.830, ANOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.17 to 0.21]
Statistical Analysis 11: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 3 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.442, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.26 to 0.11]
Statistical Analysis 12: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 3 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.358, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.11 to 0.29]
Statistical Analysis 13: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 4 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.714, ANOVA
Statistical Analysis 14: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 4 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.683, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.29 to 0.19]
Statistical Analysis 15: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 4 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.413, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.34 to 0.14]
Statistical Analysis 16: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 4 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.699, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.21 to 0.31]
Statistical Analysis 17: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 5 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.244, ANOVA
Statistical Analysis 18: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 5 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.833, ANOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-0.21 to 0.26]
Statistical Analysis 19: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 5 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.156, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.41 to 0.07]
Statistical Analysis 20: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 5 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.128, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.06 to 0.46]
Statistical Analysis 21: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 6 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.359, ANOVA
Statistical Analysis 22: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 6 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.278, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.12 to 0.43]
Statistical Analysis 23: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 6 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.699, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.33 to 0.22]
Statistical Analysis 24: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 6 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.172, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.09 to 0.50]
Statistical Analysis 25: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 7 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.515, ANOVA
Statistical Analysis 26: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 7 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.527, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.19 to 0.37]
Statistical Analysis 27: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 7 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.545, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.37 to 0.19]
Statistical Analysis 28: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 7 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.250, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.12 to 0.47]
Statistical Analysis 29: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 8 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.568, ANOVA
Statistical Analysis 30: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 8 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.381, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.16 to 0.41]
Statistical Analysis 31: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 8 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.863, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.31 to 0.26]
Statistical Analysis 32: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 8 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.330, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.16 to 0.46]
Statistical Analysis 33: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 9 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.167, ANOVA
Statistical Analysis 34: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 9 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.165, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.09 to 0.50]
Statistical Analysis 35: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 9 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.564, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.39 to 0.21]
Statistical Analysis 36: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 9 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.068, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.02 to 0.62]
Statistical Analysis 37: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 10 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.131, ANOVA
Statistical Analysis 38: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 10 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.119, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.06 to 0.56]
Statistical Analysis 39: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 10 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.616, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.39 to 0.23]
Statistical Analysis 40: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 10 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.056, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.01 to 0.66]
Statistical Analysis 41: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 11 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.255, ANOVA
Statistical Analysis 42: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 11 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.144, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.08 to 0.57]
Statistical Analysis 43: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 11 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.935, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.34 to 0.31]
Statistical Analysis 44: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 11 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.153, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.10 to 0.61]
Statistical Analysis 45: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 12 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.128, ANOVA
Statistical Analysis 46: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 12 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.067, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.02 to 0.63]
Statistical Analysis 47: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 12 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.999, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.33 to 0.33]
Statistical Analysis 48: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 12 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.088, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.05 to 0.66]
Statistical Analysis 49: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.195, ANOVA
Statistical Analysis 50: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.175, ANOVA; LS Mean Difference = 0.3, 95% CI 2-sided [-0.12 to 0.67]
Statistical Analysis 51: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.610, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.50 to 0.30]
Statistical Analysis 52: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 24 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.083, ANOVA; LS Mean Difference = 0.4, 95% CI 2-sided [-0.05 to 0.81]
Statistical Analysis 53: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 30 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.884, ANOVA
Statistical Analysis 54: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 30 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.833, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.43 to 0.35]
Statistical Analysis 55: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 30 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.620, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.49 to 0.29]
Statistical Analysis 56: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 30 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.788, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.36 to 0.48]
Statistical Analysis 57: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 36 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.755, ANOVA
Statistical Analysis 58: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 36 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.787, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.45 to 0.34]
Statistical Analysis 59: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 36 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.455, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.56 to 0.25]
Statistical Analysis 60: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 36 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.654, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.33 to 0.53]
Statistical Analysis 61: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.370, ANOVA
Statistical Analysis 62: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.472, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.51 to 0.24]
Statistical Analysis 63: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.427, ANOVA; LS Mean Difference = 0.2, 95% CI 2-sided [-0.23 to 0.53]
Statistical Analysis 64: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 48 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.159, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.69 to 0.11]
Statistical Analysis 65: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 54 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.480, ANOVA
Statistical Analysis 66: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 54 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.238, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.59 to 0.15]
Statistical Analysis 67: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 54 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.794, ANOVA; LS Mean Difference = -0.0, 95% CI 2-sided [-0.42 to 0.32]
Statistical Analysis 68: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 54 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.395, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.57 to 0.23]
Statistical Analysis 69: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 60 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.400, ANOVA
Statistical Analysis 70: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 60 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.176, ANOVA; LS Mean Difference = -0.2, 95% CI 2-sided [-0.61 to 0.11]
Statistical Analysis 71: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 60 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.573, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.47 to 0.26]
Statistical Analysis 72: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 60 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.466, ANOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-0.53 to 0.24]
Statistical Analysis 73: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.092, ANOVA
Statistical Analysis 74: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; 72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.086, ANOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-0.67 to 0.04]
Statistical Analysis 75: Comparison: Placebo Combined vs Ibuprofen Twice Daily; 72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.616, ANOVA; LS Mean Difference = 0.1, 95% CI 2-sided [-0.27 to 0.45]
Statistical Analysis 76: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; 72 Hours: Analysis was performed using an ANOVA model with treatment, baseline categorical PSR and sex terms; Test type: Superiority or Other; p = 0.040, ANOVA; LS Mean Difference = -0.4, 95% CI 2-sided [-0.79 to -0.02]

9. Secondary Outcome: Participant's Global Assessment of Medication at Day 4
Description: Participants were asked the following question: "How would you rate this medication as a pain reliever?" Participant's response was recorded using a five point scale: 1 = Very Poor, 2 = Poor, 3 = Fair, 4 = Good, 5 = Very Good, where higher score indicated better response.
Time Frame: Day 4
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 83 | 60 | 62
units on a scale | 2.3 (1.08) | 2.4 (1.15) | 2.2 (1.19)
Statistical Analysis 1: Comparison: Placebo Combined vs Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; Analysis was performed using Cochran-Mantel-Haenszel (CMH) test with modified ridit scores, controlling for baseline categorical PSR (BLPSR) and sex; Test type: Superiority or Other; p = 0.751, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo Combined vs Ibuprofen Three Times Daily; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.696, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = -0.0, 95% CI 2-sided [-0.28 to 0.20]
Statistical Analysis 3: Comparison: Placebo Combined vs Ibuprofen Twice Daily; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.760, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.0, 95% CI 2-sided [-0.21 to 0.29]
Statistical Analysis 4: Comparison: Ibuprofen Twice Daily vs Ibuprofen Three Times Daily; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.463, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = -0.1, 95% CI 2-sided [-0.36 to 0.16]

10. Secondary Outcome: Percentage of Participants Taking Rescue Medication
Description: Acetaminophen 500 milligram (mg) every 6 hours as needed was used as rescue analgesia/therapy during the course of the study.
Time Frame: Baseline up to Day 4
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 83 | 60 | 62
percentage of participants | 0 | 0 | 0

11. Secondary Outcome: Time to First Use of Rescue Medication
Description: Time to first us of rescue medication was defined as time (in hours) from a dose of study medication to the first use of recue medication and was censored at the time of the next dose of study medication, or at 12 hours after the final application of the study medication. Acetaminophen 500 milligram (mg) every 6 hours as needed was used as rescue analgesia/therapy during the course of the study.
Time Frame: Baseline up to Day 4
Population: Due to change in conduct of study no rescue medication was use, therefore data for this outcome measure was not collected and analyzed.
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Number of Doses of Rescue Medication
Description: as for outcome 10
Time Frame: Baseline up to Day 4
Population: as for outcome 11
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo Combined | Ibuprofen Twice Daily | Ibuprofen Three Times Daily
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/60 | 0/62
Other Adverse Events (participants affected / at risk) | 0/83 | 0/60 | 4/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Combined (N=83) | Ibuprofen Twice Daily (N=60) | Ibuprofen Three Times Daily (N=62)
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.